CLINICAL TRIAL: NCT00474643
Title: Correlation of Hyperghrelinemia With Carotid Artery Intima-Media Thickness in Children With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2006-06-043
Record Dates: First submitted 2007-05-10; First posted 2007-05-17 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Prader Willi Syndrome; Obesity
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prader-Willi syndrome (PWS) is a genetic disorder characterized by childhood-onset obesity and endocrine dysfunction that leads to cardiovascular disability and early death within the first 3 decades of life.To assess the significance of risk factors for future disabilities, carotid artery intima-media thickness (IMT) was measured and correlated with known atherosclerotic risk factors in 27 children with PWS and 24 age-, sex-, and body mass index (BMI)-adjusted controls.

DETAILED DESCRIPTION:
Main outcome measures: Correlation of IMT with age, standard deviation score of BMI (BMI-SDS), high-density lipoprotein cholesterol (HDL), low-density lipoprotein cholesterol (LDL), C-reactive protein, HOMA-IR and ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* Prader Willi syndrome
* Children with obesity

Exclusion Criteria:

* Acute illness
* On regular medications except growth hormone

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Hoon Paik, M.D., Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine